CLINICAL TRIAL: NCT05634226
Title: Oral Positive Pressure Device (oPEP) Effect on Flow Pulsatility in the Fontan Circuit
Brief Title: Simple Non-invasive Breathing Device to Improve Pulmonary Flow Pusatility in Single Ventricle Post Fontan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarek Alsaied (Other)
Responsible Party: Sponsor-Investigator, Tarek Alsaied, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY22050151
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Single-ventricle
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hands-free oral-positive pressure device (oPEP) (Experimental)
  Interventions: Device: Hands-free oral-positive pressure device (oPEP)

INTERVENTIONS:
Device: Hands-free oral-positive pressure device (oPEP) — This is a pilot study using a novel, minimal risk, portable, hands-free oral-positive pressure device (oPEP) in patients with Fontan palliation that will examine whether using this device in both the acute and chronic phase will alter Fontan hemodynamics and create pulsatility in the Fontan circuit and thereby increasing cardiac output. This device is easy to use and poses no significant risk to human subjects. We will measure this through echocardiographic measures including pulsatility in different aspects of the Fontan circuit including IVC, hepatic veins, the Fontan conduit, and pulmonary arteries and aortic blood flow measurements. After demonstration of how to use the device appropriately, we will have patients use the device after their clinical echocardiogram for their clinic appointment. We will ask them to use the device at home 3-4 times a day for 10-15 mins and have them return in approximately 4 weeks to have another echocardiogram done with the same measurements.

SUMMARY:
This is a pilot study using a novel, minimal risk, portable, hands-free oral-positive pressure device (oPEP) in patients with Fontan palliation that will examine whether using this device in both the acute and chronic phase will alter Fontan hemodynamics and create pulsatility in the Fontan circuit and thereby increasing cardiac output. This device is easy to use and poses no significant risk to human subjects. The investigators will measure this through echocardiographic measures including pulsatility in different aspects of the Fontan circuit including IVC, hepatic veins, the Fontan conduit, and pulmonary arteries and aortic blood flow measurements. After demonstration of how to use the device appropriately, the investigators will have patients use the device after their clinical echocardiogram for their clinic appointment. The investigators will ask them to use the device at home 3-4 times a day for 10-15 mins and have them return in approximately 4 weeks to have another echocardiogram done with the same measurements.

DETAILED DESCRIPTION:
The aortic VTI secondary outcome was inadvertently left out of the initial registration and is now reported

ELIGIBILITY:
Inclusion Criteria:

* Patients with single ventricle with Fontan palliation
* Over the age of 8 years who would be cooperative with breathing through the oPEP device

Exclusion Criteria:

* Patients with Fontan palliation under the age of 8 years
* Patients who have interrupted inferior vena cava
* Patients with abnormal pulmonary artery anatomy

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Children's Hospital Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hands-free Oral-positive Pressure Device (oPEP)
Started | 15
Completed | 11
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Hands-free Oral-positive Pressure Device (oPEP)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Pulsatility Index
Description: This will be measured by echocardiogram using Doppler evaluation of the pulmonary artery
  The Pulmonary Artery Pulsatility Index (PAPI) is calculated using Doppler-derived pulmonary artery velocities:
  PAPI= (Systolic Velocity - Diastolic Velocity) /Mean Velocity
Time Frame: The change is between enrollment echocardiogram and echocardiogram after 4 week use of the device
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Hands-free Oral-positive Pressure Device (oPEP)
Number analyzed (Participants) | 11
Ratio
  Baseline | 51.6 (16.6)
  Post treatment | 57.6 (21.1)
Statistical Analysis 1: Comparison: Hands-free Oral-positive Pressure Device (oPEP); Test type: Superiority; p = 0.1, t-test, 2 sided

2. Secondary Outcome: Aortic Valve VTI
Description: This was measured by echocardiography
  Aortic Valve Velocity Time Integral (VTI) Definition: Aortic VTI is a key echocardiographic measurement reflecting stroke distance and cardiac output.
  Measurement:
  Obtained using pulsed-wave Doppler at the left ventricular outflow tract (LVOT) just below the aortic valve.
  The VTI is measured by tracing the Doppler envelope of the LVOT flow during systole.
  Clinical Importance:
  Stroke Volume Calculation:
  Stroke Volume = LVOT VTI × LVOT Area
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Hands-free Oral-positive Pressure Device (oPEP)
Number analyzed (Participants) | 15
cm/sec
  Baseline | 19.8 (4.9)
  Post device use | 17.4 (1.8)
Statistical Analysis 1: Comparison: Hands-free Oral-positive Pressure Device (oPEP); Test type: Superiority; p = 0.06, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Hands-free Oral-positive Pressure Device (oPEP)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT05634226/Prot_SAP_001.pdf